CLINICAL TRIAL: NCT02779868
Title: Effect of Omega-3 Supplementation on Body Composition, Functional Capacity, Inflammatory Profile and Quality of Life in Cervix Cancer Patients Undergoing Chemoradiotherapy
Brief Title: Omega-3 Supplementation in Cervix Cancer Patients Undergoing Chemoradiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brazilian National Cancer Institute (Other Government)
Responsible Party: Principal Investigator, Gabriela Villaça Chaves, PhD, Researcher at Brazilian National Cancer Institute, Brazilian National Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1.150.108/2015
Record Dates: First submitted 2016-05-17; First posted 2016-05-23 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Sarcopenia
Keywords: body composition; functional capacity; quality of life
MeSH Terms: conditions — Sarcopenia | interventions — Docosahexaenoic Acids; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 (Experimental): Group who will receive 2g eicosapentaenoic (4 capsules) acid per day during the chemoradiotherapy protocol.
  Interventions: Dietary Supplement: Omega-3
- Olive oil (Placebo Comparator): Group who will receive olive oil per day (4 capsules) during the chemoradiotherapy protocol.
  Interventions: Dietary Supplement: Olive oil

INTERVENTIONS:
Dietary Supplement: Omega-3 — patients included in this group will take 2g (4 capsules) per day of eicosapentaenoic acid.
  Other Names: intervention group
  Arms: Omega-3
Dietary Supplement: Olive oil — patients included in this group will take 4 capsules per day of olive oil.
  Other Names: placebo group
  Arms: Olive oil

SUMMARY:
Cancer cachexia is a complex metabolic process affecting up to 80% of patients suffering from an advanced-stage cancer. Moreover, 20 to 40% of all cancer deaths are caused directly by cachexia. Recently, omega-3 fatty acids have gained interest for their beneficial effects in cancer cachexia. Moreover, nutritional supplementation enriched with omega-3 could potentially maintain body weight in cancer patients undergoing intensive treatment.

The investigators aims in this study is to evaluate the effect of omega-3 supplementation on body composition, functional capacity, inflammatory profile and quality of life in cervix cancer patients undergoing chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Cervix cancer at FIGO stage II and III
* Chemoradiotherapy treatment proposal (cisplatin + radiotherapy)
* Nutritional diagnosis of pre-cachexia ou cachexia

Exclusion Criteria:

* metastasis (FIGO stage IV)
* Nutritional diagnosis of refractary cachexia

Ages: 20 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in Body composition | 45 days
  Change from baseline body composition assessed by computed tomography scans before and at the end of chemotherapy treatment (45 day after the first chemotherapy)

SECONDARY OUTCOMES:
Change in Quality of life | 45 days
  Change in quality of life assessed by EORCT QL30 questionaire before and at the end of chemotherapy treatment (45 day after the first chemotherapy)
Change in Quality of life | 45 days
  Change in quality of life assessed by and EQ-5D-3L questionaire before and at the end of chemotherapy treatment (45 day after the first chemotherapy)
Change in IL-6 serum levels | 45 days
  Change in serum levels of IL-6 (ng/mL) before and at the end of chemotherapy (45 days)
Change in IL-1 serum levels | 45 days
  Change in serum levels of IL-1 (ng/mL) before and at the end of chemotherapy (45 days)
Change in TNF-alfa serum levels | 45 days
  Change in serum levels of TNF-alfa (ng/mL) before and at the end of chemotherapy (45 days)
Change in INF-gama serum levels | 45 days
  Change in serum levels of INF-gama (ng/mL) before and at the end of chemotherapy (45 days)
Change in membrane incorporation of non-esterified fatty acids | 45 days
  Change in membrane incorporation of non-esterified fatty acids assessed by Gas chromatography of fatty acid methyl esters (nmol/mL)
Change in handgrip strength | 45 days
  change in handgrip strength before and at the end of chemotherapy treatment (45 days)
Change in functional capacity (30 second stand chair test) | 45 days
  change in functional capacity assessed by 30 second stand chair test before and at the end of chemotherapy treatment (45 days)
chemoradiotherapy toxicity | 15 and 45 days
  chemoradiotherapy will be assessed by Chemotherapy toxicity criteria (CTC) version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Mariah A Aredes, Ms, Study Chair — Brazilian National Cancer Institute
Locations (1):
- Brazilian National Cancer Institute, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided